CLINICAL TRIAL: NCT00507884
Title: Pilot Study to Develop 3 Tesla MRI for Evaluation of Renal Tumors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0875
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Kidney Neoplasms
Keywords: Kidney Neoplasms; Renal Tumors; Magnetic Resonance Imaging; 3 Tesla MRI; MRI
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3 Tesla MRI: Patients with renal tumors scheduled to have a CT scan of the kidneys and abdomen.
  Interventions: Procedure: 3 Tesla MRI Scan

INTERVENTIONS:
Procedure: 3 Tesla MRI Scan — MRI of the kidneys and abdomen to be done within 15 days following the routine CT and lasting 1 - 2 hours.

SUMMARY:
The goal of this clinical research study is to find out if "3 Tesla" MRI is as good as CT scan in the evaluation of kidney tumor(s).

Objectives:

To provide preliminary data to enable subsequent development of an MRI protocol at 3 Tesla for evaluation of renal tumors and their vascular supply, which can be adopted in patients who are unable to undergo CT evaluation.

DETAILED DESCRIPTION:
"3 Tesla" MRI is a new MRI scanner that in theory, can produce better images than currently available MRI scanners.

Currently, CT scanning is the main way of evaluating tumors in the kidneys. However, there are some patients who cannot have CT scans (usually, because of allergy to CT contrast medium or kidney damage/failure). It is with these patients that researchers are hoping to use a technique (using MRI) that is as good as CT scanning.

As part of your standard of care, your doctor is requesting a CT scan of your kidneys and abdomen. If you take part in this study, you will have a "3 Tesla" MRI scan of your kidneys and abdomen as well, within 15 days following your routine CT.

For the "3 Tesla" MRI scan, you will be lying flat on the MRI scanner, and as with a regular scan, you will have a small needle placed in a vein in your arm to inject the contrast dye. A diuretic, Lasix, will be given to help distend the internal tubes in the kidney to help view your kidney better. The MRI scan will take between 1-2 hours to perform. As with regular scans, you may be asked to hold your breath on occasions.

If there is a concern about your kidney function, blood (about 1 teaspoon) will be drawn to test your kidney function before you have the MRI.

Your participation in the study will be complete at the end of the MRI scan. The routine CT scan will be the main decision making examination. However, if the MRI shows something different and potentially relevant to your care, your referring physician will be informed.

This is an investigational study. A total of 45 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone or are due to undergo a CT Renal Protocol study, in the course of pre-operative evaluation for renal tumor surgery.
2. Written informed consent will be obtained.

Exclusion Criteria:

1. Patients with an allergy to both gadopentetate dimeglumine and gadodiamide MRI contrast agents.
2. Patients with certain metallic implants, e.g., cardiac pacemakers, cardiac defibrillators, aneurysm clips, neurostimulators, and certain metallic foreign bodies. Implanted medical devices must be MRI compatible at 3.0 Tesla field strengths.
3. Patients with claustrophobia, or requiring sedation for the MRI scan.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants with renal tumors scheduled to have a CT scan of the kidneys and abdomen.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2005-03 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of CT and MRI scans of patients with renal cell carcinoma in evaluating each of nine imaging variables. | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Chaan Ng, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org